CLINICAL TRIAL: NCT04050280
Title: A Phase II Study of Cladribine, Cytarabine, and Granulocyte-Colony Stimulating Factor With Fractionated Gemtuzumab Ozogamicin (CLAG-GO) for the Treatment of Patients With Persistent, Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: CLAG-GO for Patients With Persistent, Relapsed or Refractory AML
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Hematologics, Inc (Unknown)
Responsible Party: Principal Investigator, Vu Duong, Assistant Professor of Medicine, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1946GCCC ; HP-00085334
Record Dates: First submitted 2019-07-16; First posted 2019-08-08 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia, Adult; Acute Myeloid Leukemia Recurrent; Acute Myeloid Leukemia, Relapsed, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Cladribine; Cytarabine; Granulocyte Colony-Stimulating Factor; Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CLAG-GO (Experimental): Cladribine, Cytarabine, and Granulocyte-Colony Stimulating Factor with Fractionated Gemtuzumab Ozogamicin (CLAG-GO)
  Interventions: Drug: Cladribine, Cytarabine, and Granulocyte-Colony Stimulating Factor with Fractionated Gemtuzumab Ozogamicin (CLAG-GO)

INTERVENTIONS:
Drug: Cladribine, Cytarabine, and Granulocyte-Colony Stimulating Factor with Fractionated Gemtuzumab Ozogamicin (CLAG-GO) — Induction:
  G-CSF 300 mcg subcutaneously daily on days 0-5.
  Cladribine 5 mg/m2 in normal saline given intravenously over 2 hours daily on days 1-5.
  Cytarabine 2000 mg/m2 in normal saline given intravenously over 4 hours daily on days 1-5.
  Gemtuzumab ozogamicin 3 mg/m2 intravenously over 2 hours on days 1 and 4, prior to cladribine and cytarabine.
  Consolidation:
  If CRMRD-, CR or CRi is confirmed by bone marrow biopsy and aspirate after induction chemotherapy, patients may receive one cycle of consolidation chemotherapy (at the discretion of the investigator) with the same CLAG-GO regimen at the same doses given for induction. In addition, the investigator has the option of giving CLAG alone without GO if there is concern for increased risk of sinusoidal obstruction syndrome.
  Patients who remain in CRMRD-, CR or CRi after consolidation chemotherapy may receive up to eight infusions of GO 2 mg/m2 approximately every 28 days.
  Other Names: Mylotarg

SUMMARY:
This study involves evaluating a combination of chemotherapy drugs known as "CLAG-GO" [cladribine, cytarabine, granulocyte-colony stimulating factor (G-CSF) and gemtuzumab ozogamicin (GO)] in the treatment of acute myeloid leukemia (AML) that has not responded well to standard therapy or has returned after an initial remission (relapsed). The trial will be conducted at the University of Maryland Greenebaum Comprehensive Cancer Center (UMGCCC). Potential participants will go through a screening period to see if they are eligible to join the study. If eligible, participants will be hospitalized for 4-5 weeks to receive study treatment with CLAG-GO, called induction chemotherapy. If tests show that the cancer is in remission after induction chemotherapy, participants may undergo further chemotherapy (known as consolidation) or may proceed with bone marrow/stem cell transplantation. Patients who receive consolidation chemotherapy and remain in remission may have up to 8 cycles of outpatient maintenance therapy. A cycle lasts about 28 days. All participants will be monitored carefully for both side effects and to see if the study treatment is working. Lab tests and exams will be conducted throughout the entire study. In addition, special studies will be done at various time points to try to understand better how the drugs work and which patients are likely to respond best.

DETAILED DESCRIPTION:
This is a single-arm, two-stage phase II trial of cladribine, cytarabine, granulocyte colony stimulating factor and gemtuzumab ozogamicin (CLAG-GO) in adult patients with acute myeloid leukemia (AML) who are either have persistent disease after initial induction chemotherapy or are in first relapse, with early stopping for unacceptable toxicity. The trial will be conducted at the University of Maryland Greenebaum Comprehensive Cancer Center (UMGCCC), with a target enrollment of 39 patients if the trial proceeds to the second stage. Eligible patients will receive induction chemotherapy with CLAG-GO at the doses detailed below. In the first stage of the trial, a sequential boundary is used to monitor induction mortality and halt accrual if this mortality is significantly above 10%. If more than 6 responses are seen in the initial 19 patients, 20 additional patients will be enrolled in the 2nd stage. Responders may proceed to allogeneic hematopoietic stem cell transplantation (alloHSCT) at any time after induction, and these patients will be monitored for at least 30 days post-transplantation for veno-occlusive disease. Responding patients will also have the option of having a single cycle of consolidation therapy using the same CLAG-GO regimen, followed by maintenance with GO monotherapy for up to 8 additional cycles. Responses will be categorized according to the European LeukemiaNet (ELN) response criteria for AML. Assessment of measureable residual disease (MRD) will be conducted with bone marrow aspirate samples and changes in immunophenotype will be evaluated. In addition, single nucleotide polymorphism (SNP) analysis and sialylation status of CD33, along with sialidase activity of myeloblasts will be evaluated and correlated with responses and survival times. Safety and toxicity will be evaluated continuously, and event-free survival, and overall survival as well as the proportion of patients proceeding to receive alloHSCT will be estimated.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients age 18 years or older, with a pathologically confirmed diagnosis of AML [excluding acute promyelocytic leukemia (APL)] according to WHO criteria. AML may be de novo, or following a prior hematologic disease and/or therapy-related.
2. Patients must have relapsed after or be refractory to at least one course of an intensive chemotherapy regimen, for example anthracycline/cytarabine ("7+3" or daunorubicin and cytarabine liposome). Patients with residual disease on day 13-22 of initial induction chemotherapy are eligible, provided the bone marrow cellularity is ≥ 30% AND bone marrow blasts are ≥ 20%. Hypomethylating agents such as azacitidine or decitabine are allowed as a prior therapy, but are not considered an intensive chemotherapy regimen.
3. Eastern Cooperative Oncology Group performance status of 0-2.
4. Any systemic chemotherapy and any radiotherapy must be completed at least 7 days prior to initiation of protocol therapy, with the exception of hydroxyurea or 6-mercaptopurine for cytoreduction.
5. At least 20% expression of CD33 as determined by flow cytometry or immunohistochemical staining.
6. Adequate renal function, defined as a serum creatinine less than 1.8 mg/dL.
7. Adequate hepatic function, defined as a direct bilirubin less than 2 times the institutional upper limit of normal (ULN) and AST, ALT and Alkaline Phosphatase less than 3 times the ULN.
8. Patients who relapse after allogeneic hematopoietic stem cell transplantation are eligible, provided they are at least 60 days from stem cell infusion, do not have > grade 1 graft versus host disease, and have been off all immunosuppressive therapy for at least 2 weeks.
9. Female patients of childbearing potential must have a negative pregnancy test and agree to use an adequate method of contraception as defined by the protocol. This must persist through the treatment period until at least 6 months after the last dose of chemotherapy or GO.
10. Male subjects who are able to father children and are having intercourse with females of childbearing potential must also agree to an acceptable method of contraception through the treatment period until at least 3 months after the last dose of chemotherapy or GO, and must refrain from sperm donation during this period.
11. Ability to give written informed consent.

Exclusion Criteria:

1. Patients with acute promyelocytic leukemia (FAB-M3) or chronic myelogenous leukemia in blast phase.
2. Isolated myeloid sarcoma. Patients must have marrow involvement with AML to enter the study.
3. Patients with known active AML involvement of the central nervous system.
4. Prior treatment with gemtuzumab ozogamicin or cladribine for AML. Prior treatment with cytarabine is permitted.
5. As patients will be receiving G-CSF prior to chemotherapy, patients presenting with symptomatic leukostasis (as judged by the investigator) are excluded. Hydroxyurea, 6-mercaptopurine and/or leukapheresis for blast count control (see inclusion criterion #4) for patients with asymptomatic hyperleukocytosis is permitted before starting treatment, but must be stopped for at least 24 hours prior to starting protocol treatment.
6. Active uncontrolled infection. Patients on prophylactic antibacterial, antifungal, and/or antiviral agents and patients whose infections are controlled with these agents are eligible.
7. Known active hepatitis B or C or other known active hepatic disorder.
8. Any history of veno-occlusive disease (VOD)/sinusoidal obstruction syndrome (SOS).
9. Active concurrent malignancy, unless disease-free for at least 3 years. Subjects with treated non-melanoma skin cancer, in situ carcinoma or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed. Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease are eligible if hormonal therapy has been initiated or the malignancy has been treated surgically or with definitive radiotherapy.
10. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that per investigator's judgment would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Response Rate (Efficacy) | Responses will be assessed following induction chemotherapy, within 14 days of documented full blood count recovery.
  Responses will be judged according to modified European LeukemiaNet recommendations published in 2017. Patients who achieve either 1) complete remission without minimal residual disease, 2) complete remission, or 3) complete remission with incomplete hematologic recovery will be considered responders
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | From date of enrollment until death from any cause, whichever comes first, assessed up to 1 year.
  All adverse events will be graded according to CTCAE version 5.

SECONDARY OUTCOMES:
Presence of minimal residual disease | Assessed at the end of induction, consolidation and maintenance therapy, up to 1 year
  This is determined by flow cytometry completed through Hematologics, Inc.
Time to relapse or death | measured from the date of confirmed remission until the date of confirmed relapse, assessed up to 2 years. Time to death (survival) is measured from the date of enrollment until the date of death, assessed up to 2 years.
  Time to relapse is measured from the date of confirmed remission until the date of confirmed relapse. Time to death (survival) is measured from the date of enrollment until the date of death, assessed up to 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Vu H. Duong, MD, MS, Principal Investigator — University of Maryland Greenebaumn Comprehensive Cancer Center
Locations (1):
- University of Maryland Greenebaumn Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Individual results will not be shared with participants nor their primary care physician. IPD (Individual Patient Data) would only be shared with the applicable regulatory parties in the event of an audit or for monitoring purposes. All HIPAA laws will be followed. We will not be sharing IPD in publications nor with other researchers not specified in the protocol. Aggregate findings will be reported in scholarly journals.